CLINICAL TRIAL: NCT05027633
Title: Immunotherapy With Chemotherapy and Chemoradiation for Advanced Squamous Cancer of Nasal Cavity / Paranasal Sinuses (I-NAPA)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-1109; NCI-2021-09409 (Other: NCI-CTRP Clinical Trials Reporting Registry)
Record Dates: First submitted 2021-08-24; First posted 2021-08-30 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Squamous Cell Carcinoma; the Nasal Cavity; Paranasal Sinuses
MeSH Terms: conditions — Carcinoma, Squamous Cell | interventions — pembrolizumab; Docetaxel; Cisplatin; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- pembrolizumab, docetaxel, and cisplatin or carboplatin (Other): IV
  Interventions: Drug: Pembrolizumab; Drug: Docetaxel; Drug: Cisplatin; Drug: Carboplatin

INTERVENTIONS:
Drug: Pembrolizumab — given by IV
Drug: Docetaxel — given by IV
Drug: Cisplatin — given by IV
Drug: Carboplatin — given by IV

SUMMARY:
This is a single arm phase II study that will evaluate the combination of pembrolizumab, docetaxel, and cisplatin or carboplatin (PDC) as single treatment modality in patients with stage II-IVb (T2-4, any N, M0) squamous cell carcinoma of the nasal cavity/paranasal sinuses (PNS SCC).

DETAILED DESCRIPTION:
Primary Objective

-Increase overall response rate (ORR), following pembrolizumab combined with induction chemotherapy prior to radiation, from historical 60% with induction chemotherapy alone to 80%.

Secondary Objective

* Improve the following efficacy endpoints relative to historical results with chemotherapy alone: progression free survival (PFS), overall survival (OS), organ [orbital, maxillary, cranial] preservation rate (OPR), and locoregional failure (LRF).
* To determine safety and tolerability of pembrolizumab combined with induction chemotherapy and chemoradiation in patients with PNS SCC.
* Correlate immune phenotype in tumors and blood, including T cell infiltration and PD-L1 status, with treatment outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Male/female participants who are at least 18 years of age on the day of signing informed consent with newly diagnosed, previously untreated, histologically and/or cytologically confirmed diagnosis of Stage II-IVb PNS SCC will be enrolled in this study.
* Male participants:

A male participant must agree to use a contraception as detailed in Appendix 3 of this protocol during the treatment period and for at least 150 days after the last dose of study treatment and refrain from donating sperm during this period.

-Female participants:

A female participant is eligible to participate if she is not pregnant (see Appendix 3), not breastfeeding, and at least one of the following conditions applies:

1. Not a woman of childbearing potential (WOCBP) as defined in Appendix 3 OR
2. A WOCBP who agrees to follow the contraceptive guidance in Appendix 3 during the treatment period and for at least 150 days after the last dose of study treatment.

   * The participant (or legally acceptable representative if applicable) provides written informed consent for the trial.
   * Have measurable disease based on RECIST 1.1.
   * Have provided archival tumor tissue sample or newly obtained core or excisional biopsy of a tumor lesion not previously irradiated. Formalin-fixed, paraffin embedded (FFPE) tissue blocks are preferred to slides. Newly obtained biopsies are preferred to archived tissue.
   * Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1. Have adequate organ function as defined in the following table (Table 1). Blood must be collected within 14 days prior to the start of study treatment.

Exclusion Criteria:

* A WOCBP who has a positive urine pregnancy test within 72 hours prior to treatment (see Appendix 3). If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti PD L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX 40, CD137).
* Patients must not have received prior systemic anti-cancer therapy including investigational agents or radiation therapy for PNS SCC but could have received treatment for prior cancers if greater than 2 years (refer to Item 8 for further details).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2021-11-02 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
To increase overall response rate (ORR) | through study completion, an average of 1 year

SECONDARY OUTCOMES:
To improve the following efficacy endpoints relative to historical results with chemotherapy alone | through study completion, an average of 1 year
To determine the safety of pembrolizumab combined with induction chemotherapy and chemoradiation in patients with PNS SCC | through study completion, an average of 1 year
To determine the tolerability of pembrolizumab combined with induction chemotherapy and chemoradiation in patients with PNS SCC | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Renata Ferrarotto, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org